CLINICAL TRIAL: NCT01587014
Title: Safety and Feasibility of Prima-Temp Thermometer Patch in Determining Baseline Temperatures of Research Subjects in a Hospital Intensive Care Unit (ICU)
Brief Title: Safety and Feasibility of Prima-Temp Thermometer Patch
Acronym: Prima-Temp
Status: Completed | Type: Observational
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Julie Dunn, M.D., Principal Investigator, Poudre Valley Health System
Other Study IDs: 1-001
Record Dates: First submitted 2012-03-01; First posted 2012-04-27 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Erythema; Edema; Papules White; Eruption
MeSH Terms: conditions — Erythema; Edema; Exanthema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test the safety and feasibility of the Prima-Temp Thermometer Patch in determining baseline temperatures of research subjects in a hospital intensive care unit (ICU).

Primary Objective: Assess safety of the Prima-Temp temperature patch with nursing staff skin site assessments.

Secondary Objective: Establish individual subject baseline temperature using intermittent temperature measurements (every 5 minutes) with the Prima-Temp thermometer patch and wireless transmission of the data to a receiver box and HIPAA compliant, centrally located personal computer (PC) and compare research subject's baseline temperature with temperatures taken in the ICU in the normal course of care.

DETAILED DESCRIPTION:
The manifestation of fever and its characteristics is essential to the care of intensive care unit patients. As a marker for infection or other disease process, the presence of a fever and its temperature peak must be reliably obtained in ICU patients and must be monitored closely to optimize effective therapy. Inherent variability of different temperature measurement methods can lead to a difficulty in determining the optimal timing of medical interventions. Ideally, nurses and medical staff in acute care hospital facilities could have a temperature monitoring system that aids recognition of fever and systemic infection that is not labor intensive and provides consistent and reliable temperatures. Automatic transmission to a data recorder lessens the chances of manual entry error into the medical record. Frequent measurements allow establishment of a patient's individual baseline temperature to provide individualized guidelines for medical interventions with an increase of 2°F above baseline as documentation of a fever. Finally, the frequent temperature monitoring should be minimally invasive and comfortable to the patient.

ELIGIBILITY:
Inclusion Criteria

1. Men and women of any race.
2. Men of age > 18 years
3. Women with no childbearing potential (age > 50, age ≥ 18 s/p hysterectomy)
4. Arm circumference >23 cm and < 38 cm

Exclusion Criteria

1. Patient with known or documented adhesive, Tegaderm allergies.
2. Abnormal axillary integument such as rashes, burns, laceration.
3. Hidradenitis suppurativa and/or dermatologic diseases that might interfere with the evaluation of the test site reactions.
4. Non-English speakers
5. Pregnant women
6. Patient requiring hypothermic therapy, with the exception of non-steroidal anti-inflammatory treatment (acetaminophen, ibuprofen, aspirin, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in hospital intensive care unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dunn, M.D., Principal Investigator — Poudre Valley Health System
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research Site Website — http://pvhs.org/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Prima-Temp Monitoring Patch: ICU patients receive the Prima-Temp Temperature Monitoring Patch.
Period: Overall Study
Arm/Group | Prima-Temp Monitoring Patch
Started | 26
Completed | 24
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: ICU patients
Groups:
- Device Arm: ICU patients receive the Prima-Temp Temperature Monitoring Patch.
Arm/Group | Device Arm
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 80]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events Experienced by Participants Between Day 0 and Day 14 After Receiving the Prima-Temp Temparature Patch
Description: The nursing staff will complete a thermometer skin site assessment daily. If the patch is removed or dislodged prior to study day 7 and 14 data points for any reason other than temporary transfer from the floor for a medical study, the nursing staff will be asked to complete an additional comfort skin site assessment. The area evaluated by the nurse will include skin in contact with both the Covidien/Kendall Lifetrace® belt and the thermometer patch.
Time Frame: 0-14 days
Measure: Number; unit: Adverse event
Arm/Group | Device Arm
Number analyzed (Participants) | 26
Adverse event | 1

2. Secondary Outcome: Determine Research Subject's Baseline Temperature.
Description: Using intermittent temperature data obtained with Prima-Temp temperature patch and wireless transmission to a receiver box and PC, researchers will compare research subject's baseline temperature with temperatures taken in the ICU in the normal course of care.
Time Frame: 0-14 days
Measure: Number; unit: data unavailable
Arm/Group | Device Arm
Number analyzed (Participants) | 26
data unavailable | 0

ADVERSE EVENTS:
Time Frame: Every 24 hours until patient was discharged from hospital, an average of 1 week
Description: Adverse events were recorded every 24 hours.
Arm/Group | Device Arm
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Arm (N=26)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No